CLINICAL TRIAL: NCT04016233
Title: A Phase I, Open-label Multiple Dose Safety, Pharmacokinetic, Pharmacodynamic, and Acceptability Study of Tenofovir Rectal Douche
Brief Title: Tenofovir Rectal Douche to Prevent HIV Transmission
Acronym: DREAM-03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00196310; 5U19AI113127 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: HIV/AIDS; HIV Prevention
Keywords: Tenofovir; Tenofovir douche
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Three TFV Medicated Douche Sequences (Experimental): Once enrolled, participants will complete a baseline sampling session and then three sequences of study product administration, each with 3 douches. Sequence A will be 3 sequential doses of TFV douche; Sequence B will be one dose of TFV douche followed by 2 sequential non-medicated douches; Sequence C will be 2 sequential non-medicated douches followed by a single dose of TFV douche. There will be a washout period of at least 14 days between sequences. Participants will have sequences administered in clinic or a research unit, followed by various specimen collections over 8 days according to individual sampling schedule assigned to each participant. Specimens will be collected on Days 1, 2, 4, and 8 post sequence administration.
  Interventions: Drug: Tenofovir douche

INTERVENTIONS:
Drug: Tenofovir douche — 660 mg TFV in 125 mL hypo-osmolar solution

SUMMARY:
DREAM-03 is an early phase-1, open label study to compare the safety, pharmacokinetics (PK), pharmacodynamics (PD), and acceptability of 3 sequences of tenofovir (TFV) and non-medicated douches. The overall goal is to inform the design of an extended safety study of an on-demand and behaviorally congruent TFV douche to confer protection from HIV acquisition in an outpatient pre-RAI context.

DETAILED DESCRIPTION:
On demand and behaviorally-congruent forms of HIV pre-exposure prophylaxis (PrEP) have long been demanded by communities at great risk of HIV, especially men who have sex with men (MSM). The DREAM Program is developing a tenofovir (TFV) douche for on demand PrEP use prior to receptive anal intercourse (RAI), given that the vast majority of MSM very commonly douche prior to RAI (behaviorally-congruent). DREAM-01 established a range of safe and acceptable TFV rectal douche formulations administered as a single dose which also achieved desired tissue concentrations of drug. DREAM Behavioral Survey data established that a series of 3 cleansing douches are typical prior to RAI in MSM.

To more closely simulate actual douching practice prior to RAI, the investigators propose the study of 3 douche product sequences to approximate the highest (3 TFV douches [Sequence A]) and lowest (only one TFV douche at the beginning [Sequence B] or end [Sequence C] of 2 other non-medicated douches) number of TFV doses in a typical repeated cleansing douche sequence. Study objectives including safety, pharmacokinetics (PK), pharmacodynamics (PD), and acceptability of repeated douching with TFV and non-medicated solutions, are essential to inform the design of an extended safety study of a TFV douche in outpatient pre-RAI contexts.

DREAM-03 is an early phase 1, open label study to compare the safety, PK, PD, and acceptability of 3 sequences of TFV and non-medicated douches. Each participant will undergo a Screening Visit to evaluate eligibility. Baseline Visit will assess pre-dose safety, PK, PD, and behavioral points of reference. Three sequences described above (Sequences A, B, and C) occur sequentially within each subject. Safety, PK, PD, and behavioral readouts are assessed at specified times over 8 hours after each dose, followed by a minimum 14 day washout period before the next sequence.

The TFV douche to be used, previously known as Product C from the DREAM-01 study, consists of TFV 660 mg in 125 mL half-normal saline (TFV 5.28 mg/mL). Sequence A includes 3 TFV douches and sequence B and C include only one TFV douche at the beginning or the end, respectively. In sequence B and C the other douches (2 per sequence) will be non-medicated solutions (tap water). Sequence A, proportional accumulation of all 3 TFV douches, would represent a 3-fold increase in TFV dose relative to the highest single dose used in DREAM-01 (Product C, 660 mg/125 mL half-normal saline [TFV 5.28 mg/mL]). Sequence B and C, with only 1 TFV douche dose either preceded by or following two non-medicated douches, are expected to exceed the tissue exposure of the lowest dose used in DREAM-01 (Product A, TFV 220 mg/125 mL normal saline).

Participant accrual will take approximately 6 months and each participant will be on study for approximately 6 months. Total study duration is about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at screening
* Willing and able to communicate in English
* Willing and able to provide written informed consent to take part in the study; non-literate individuals may indicate consent with a thumbprint accompanied by the signature of an objective witness
* Willing and able to provide adequate locator information
* Understand and agree to local Sexually Transmitted Infection (STI) reporting requirements
* HIV-1 uninfected at screening as documented by Combo Ag/Ab HIV-1/HIV-2 immunoassay (refer to Appendix II for confirmatory testing algorithm)
* Available to return for all study visits, barring unforeseen circumstances
* Per participant report at screening, a history of consensual Receptive Anal Intercourse (RAI) at least five times in lifetime
* Per participant report at screening, experience with receiving or self-administering multiple rectal douches in the context of RAI in the past year.
* If the study participant is currently prescribed oral Tenofovir Disoproxil Fumarate (TDF) 300 mg/Emtricitabine (FTC) 200 mg (TruvadaTM) as HIV Pre-Exposure Prophylaxis (PrEP), the participant may continue to take oral TDF/FTC as prescribed as long as the participant agrees to adhere to a consistent dosing schedule throughout the study duration.
* If of reproductive potential (defined as pre-menopausal cisgender women or transgender men who have not had a sterilization procedure per self-report, such as hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy), must have a negative beta human chorionic gonadotropin (βHCG) pregnancy test (sensitivity of ≤ 25 milli-international units per milliliter (mIU/mL)) performed (and results known) on the same day as and before initiating the protocol-specified study product at Visit 3.
* If of reproductive potential, women must agree to use a reliable form of contraception, during the trial and for 4 weeks after the final study product doses, from the list below:

  1. Intrauterine device (IUD) or intrauterine system (IUS) that meets <1% failure rate as stated in the product label.
  2. Hormone-based contraceptive that meets <1% failure rate as stated in the product label
* Willing to abstain from insertion of anything (drug/medication, penis, object, sex toy, or douche) into the anorectum for 72 hours before and after each research unit study product exposure and 7 days after each flexible sigmoidoscopy with biopsy collection.
* Willing to refrain from aspirin and Nonsteroidal anti-inflammatory drug (NSAID) use for one week before and after each study biopsy visit
* Willing and able to use condoms provided by the study for all RAI for the duration of participation
* Agrees not to participate in other research studies involving drugs and/ or medical devices for the duration of the study

Exclusion Criteria:

* History of Hepatitis B infection, as documented by positive HBsAg at screening
* ≥ Grade 2 laboratory abnormality at baseline as defined by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 - July 2017, and Addendum 3 (Rectal Grading Tables for Use in Microbicide Studies)
* Significant colorectal symptom(s) as determined by medical history or by participant self-report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
* At screening or within the past 2 months: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active Herpes Simplex Virus (HSV) lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts. Note that HSV seropositivity with no active genital lesions is not an exclusion criterion. (Note: if an STI apart from HIV is detected, the participant will be referred for treatment and can be retested in 30 days and rescreened once.)
* History of an underlying clinically significant cardiac arrhythmia or renal disease (including creatinine clearance <60 mL/min using Cockcroft-Gault equation)
* Serum phosphate < 2.3 mg/dL
* History of severe or recent cardiac or pulmonary event
* History of significant gastrointestinal bleeding
* Current use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], NSAIDs, or Pradaxa®)
* Use of systemic or anorectal immunomodulatory medications within 4 weeks of enrollment or planned use at any time during study participation
* Per participant report, use of any rectally administered products containing N-9 (including condoms) or investigational products within 4 weeks of enrollment, or planned use of either at any time during study participation
* Known allergic reaction to TFV or other components of the test articles
* Current known HIV-infected partner(s)
* History of recurrent urticaria
* Symptoms suggestive of acute HIV seroconversion at screening and enrollment
* Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Change in Tenofovir Diphosphate (TFV-DP) concentration | At 1 hour, 3 hours, 6 hours, 24 hours, 72 hours, 168 hours after each TFV douche sequence administration
  Colonic tissue cell TFV-DP concentrations (femtomoles/million cells) will be measured after each study douche sequence administration, based on the individual participant's sampling schedule, on Day 1 (at 1 hour, 3 hours, or 6 hours post dose), Day 2 (24 hours post dose), Day 4 (72 hours post dose), or Day 8 (168 hours post dose).
Acceptability of TFV Douche Sequence A as assessed by Sequence A Acceptability Questionnaire | Following administration of study product sequence A, up to 1 hour
  To analyze study product sequence acceptability, the outcome will be examined in both continuous and dichotomous forms. For each sequence, descriptive statistics of overall acceptability will be generated (i.e., mean and standard deviation for continuous variables and proportion of subjects who consider the sequences acceptable -- with score 3 or greater). The acceptability of each sequence is defined as a mean score of 3 on 4-point continuous acceptability measure (1=completely unacceptable; 2=somewhat unacceptable; 3=somewhat acceptable; 4=highly acceptable) that is defined in this study as the minimal clinically meaningful threshold for sequence acceptability. Each sequence acceptability questionnaire consists of 6 sections with 36 questions total.
Acceptability of TFV Douche Sequence B as assessed by Sequence B Acceptability Questionnaire | Following administration of study product sequence B, up to 1 hour
  To analyze study product sequence acceptability, the outcome will be examined in both continuous and dichotomous forms. For each sequence, descriptive statistics of overall acceptability will be generated (i.e., mean and standard deviation for continuous variables and proportion of subjects who consider the sequences acceptable -- with score 3 or greater). The acceptability of each sequence is defined as a mean score of 3 on 4-point continuous acceptability measure (1=completely unacceptable; 2=somewhat unacceptable; 3=somewhat acceptable; 4=highly acceptable) that is defined in this study as the minimal clinically meaningful threshold for sequence acceptability. Each sequence acceptability questionnaire consists of 6 sections with 36 questions total.
Acceptability of TFV Douche Sequence C as assessed by Sequence C Acceptability Questionnaire | Following administration of study product sequence C, up to 1 hour
  To analyze study product sequence acceptability, the outcome will be examined in both continuous and dichotomous forms. For each sequence, descriptive statistics of overall acceptability will be generated (i.e., mean and standard deviation for continuous variables and proportion of subjects who consider the sequences acceptable -- with score 3 or greater). The acceptability of each sequence is defined as a mean score of 3 on 4-point continuous acceptability measure (1=completely unacceptable; 2=somewhat unacceptable; 3=somewhat acceptable; 4=highly acceptable) that is defined in this study as the minimal clinically meaningful threshold for sequence acceptability. Each sequence acceptability questionnaire consists of 6 sections with 36 questions total.
Change in participant behavior from baseline and study product desirability as assessed by In-Depth Interview | Upon completion of the study at final visit, up to 2 hours
  A final In-depth Interview will be conducted over the telephone by a trained interviewer. This interview will explore associations between baseline behavior, experience using the products during the study, and likelihood of product use in the future. This interview will take place at the final clinic visit after all behavioral assessments have been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No